CLINICAL TRIAL: NCT03061825
Title: Post-Market Study for Zenith Alpha™ Abdominal Endovascular Graft
Brief Title: Zenith Alpha™ Abdominal Endovascular Graft
Status: Completed | Type: Observational
Sponsor: Cook Research Incorporated (Industry)
Responsible Party: Sponsor
Organization: Cook Group Incorporated (Industry)
Other Study IDs: 15-10
Record Dates: First submitted 2017-02-20; First posted 2017-02-23 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Abdominal Aortic; Aorto-iliac Aneurysm
Keywords: Aneurysm; Aortic Aneurysm; Aortic Aneurysm, Abdominal; Iliac Aneurysm; Vascular Diseases; Cardiovascular Diseases; Aortic Diseases
MeSH Terms: conditions — Aneurysm; Aortic Aneurysm; Aortic Aneurysm, Abdominal; Iliac Aneurysm; Vascular Diseases; Cardiovascular Diseases; Aortic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Zenith Alpha™ Abdominal Endovascular Graft — Zenith Alpha™ Abdominal Endovascular Graft for the treatment of abdominal aortic or aorto-iliac aneurysm.

SUMMARY:
The purpose of this study is to evaluate the clinical performance of the Zenith Alpha™ Abdominal Endovascular Graft for the treatment of abdominal aortic or aorto-iliac aneurysm.

ELIGIBILITY:
Inclusion Criteria:

* A patient is considered eligible for inclusion in the study if the patient has an infrarenal abdominal aortic or aorto-iliac aneurysm and is intended to be treated with the Zenith Alpha™ Abdominal Endovascular Graft

Exclusion Criteria:

* Life expectancy less than (<) 2 years
* Inability or refusal to give informed consent by the patient or legally authorized representative
* Unwilling or unable to comply with the study follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential study patients with abdominal aortic or aorto-iliac aneurysm will be "screened " at the hospital.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2021-01-06 (Actual); Study Completion 2021-01-06 (Actual)

PRIMARY OUTCOMES:
Device Success | 2 years
  Technical success (successful introduction and deployment of the device in the absence of surgical conversion or mortality) plus freedom from the following: abdominal aneurysm rupture, conversion, Type I or III endoleak, graft limb occlusion and abdominal aneurysm size increase > 5 mm.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Forbes, MD, Principal Investigator — Toronto General Hospital
Locations (5):
- Canada (5):
  - Vancouver Hospital and Health Science Center, Vancouver, British Columbia
  - Nova Soctia Health Authority, Halifax, Nova Scotia
  - Hamilton General Hospital, Hamilton, Ontario
  - London Health Sciences Center, London, Ontario
  - Toronto General Hospital, Toronto, Ontario